CLINICAL TRIAL: NCT05998135
Title: Phase II Clinical Trial Repurposing Atovaquone for the Treatment of Platinum-Resistant Ovarian Cancer
Brief Title: Repurposing Atovaquone for the Treatment of Platinum-Resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Namita Khanna, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005363; NCI-2023-03479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00005363 (Other: Emory University); WINSHIP5782-22 (Other: Emory University); P30CA138292 (NIH)
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Ovarian High Grade Serous Adenocarcinoma; Platinum-Resistant Ovarian Carcinoma
MeSH Terms: interventions — Atovaquone; Biopsy; Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (atovaquone) (Experimental): Patients receive atovaquone PO on study. Patients also undergo CT and biopsy or paracentesis throughout the study.
  Interventions: Drug: Atovaquone; Procedure: Biopsy; Procedure: Computed Tomography; Procedure: Paracentesis

INTERVENTIONS:
Drug: Atovaquone — Given PO
  Other Names: 566C80; BW-566C; BW-A566C; Mepron
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Paracentesis — Undergo paracentesis

SUMMARY:
This phase II trial test tests how well repurposing atovaquone works in treating patients with platinum-resistant ovarian cancer. Atovaquone is used for the treatment or prevention of certain infections. Atovaquone is in a class of medications called antiprotozoal agents. It works by stopping the growth of certain types of protozoa that can cause pneumonia. Giving atovaquone may be effective in treating platinum-resistant ovarian cancer and result in improved outcomes compared to standard chemotherapy regimens.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine progression free survival of twenty-eight patients with platinum-resistant ovarian cancer treated with atovaquone.

SECONDARY OBJECTIVES:

I. To determine clinical benefit rate (complete response, partial response or stable disease) at six months.

II. To determine overall survival. III. To quantitate the on-target STAT3 inhibitory effect of atovaquone on STAT3-dependent gene transcription.

IV. To quantitate changes of the tumor immune infiltrate by inhibition of STAT3 with atovaquone.

OUTLINE:

Patients receive atovaquone orally (PO) on study. Patients also undergo computed tomography (CT) and biopsy or paracentesis throughout the study.

After completion of study treatment, patients are followed up for 30 days and then every 6 month thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with platinum-resistant, high-grade serous ovarian cancer, defined as disease progression within six months of completion of their last platinum-based chemotherapy
* Patients must maintain Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* There will be no limitations on number of prior lines of therapy
* Trial is open to non-English speaking patients
* Trial is open to patients referred from community practice

Exclusion Criteria:

* Patients who are < 18 years old
* Patients who are pregnant or breastfeeding (due to cancer of their reproductive organs, patients enrolled in the trial are unable to conceive)
* Patients who are incarcerated
* Patients who are unable to provide consent / lack decision-making capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From initiation of atovaquone to progression or death, assessed up to 1 year
  Will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median PFS will be estimated using the Brookmeyer-Crowley approach.

SECONDARY OUTCOMES:
Clinical benefit rate | At 6 months
  Clinical benefit rate is defined as complete response, partial response, and/or stable disease at six months. Clinical response will be assessed every 6 weeks for the first 24 months and every 12 weeks thereafter using Response Evaluation Criteria in Solid Tumors 1.1 criteria. Will be estimated as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method.
Overall survival (OS) | From diagnosis to death from any cause, where patients who are alive will be censored at last follow-up date, assessed up to 1 year
  OS will be estimated using the Kaplan-Meier method, and median survival will be calculated. A 95% confidence interval will be estimated using the Brookmeyer-Crowley approach.
Incidence of adverse events | Up to 30 days
  Safety will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. Frequencies and percentages will be used to summarize safety events.

CONTACTS AND LOCATIONS:
Overall Officials: Namita Khanna, MD, MSPH, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States